CLINICAL TRIAL: NCT06999044
Title: Study on the Optimization of the Diagnostic Process for Chronic Rhinitis Using Nasal Allergen Provocation Test
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-SR-1114
Record Dates: First submitted 2025-04-07; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Chronic Rhinitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- chronic rhinitis: The examination room temperature was maintained at 20-22°C, with patients acclimatizing to the testing environment for 15-30 minutes prior to evaluation. Baseline assessments included 4-phase rhinomanometry (4PR) and subjective symptom evaluation using a visual analogue scale (VAS) and total nasal symptom scores (TNSS). A reagent devoid of dust mite allergen was applied to the mucosa above the inferior nasal turbinate (middle meatus side) or the medial surface. After a 15-minute observation period, the test was terminated if a positive reaction occurred.
  If no positive reaction was observed, formal graded-concentration testing commenced. Starting with the predefined lowest concentration, patients were monitored for 15 minutes. A positive reaction prompted immediate termination of the test, followed by nasal secretion collection, reassessment of subjective/objective parameters, data recording, and administration of sychallenge protocols and ARIA guideline criteria for symptom scoring.
- Healthy Volunteers: The examination room temperature was maintained at 20-22°C, with patients acclimatizing to the testing environment for 15-30 minutes prior to evaluation. Baseline assessments included 4-phase rhinomanometry (4PR) and subjective symptom evaluation using a visual analogue scale (VAS) and total nasal symptom scores (TNSS). A reagent devoid of dust mite allergen was applied to the mucosa above the inferior nasal turbinate (middle meatus side) or the medial surface. After a 15-minute observation period, the test was terminated if a positive reaction occurred.
  If no positive reaction was observed, formal graded-concentration testing commenced. Starting with the predefined lowest concentration, patients were monitored for 15 minutes. A positive reaction prompted immediate termination of the test, followed by nasal secretion collection, reassessment of subjective/objective parameters, data recording, and administration of symptomatic relief medication. Absence of reactivity triggered progres

SUMMARY:
Chronic rhinitis (CR) is one of the most prevalent global diseases, with studies estimating that up to 30% of the worldwide population is affected. In China, the prevalence of chronic rhinitis ranges from 10% to 40%, impacting over 300 million individuals. Although non-fatal, CR significantly disrupts daily work and academic performance, predisposes patients to respiratory comorbidities such as nasal polyps and asthma, and may induce systemic complications (e.g., secretory otitis media). Additionally, it detrimentally affects mental health, contributing to psychological disorders, substantial healthcare expenditures, and socioeconomic burdens.

Clinically, CR is broadly classified into allergic rhinitis (AR) and non-allergic rhinitis (NAR) based on skin prick test (SPT) and/or serum-specific IgE results. However, real-world clinical complexity arises as a subset of patients exhibit AR symptoms despite negative test results (local allergic rhinitis), while others with confirmed AR evade detection via conventional methods. This challenges the traditional dichotomous classification, highlighting its growing inadequacy. Given divergent therapeutic strategies for CR subtypes, ambiguous classification frequently leads to ineffective clinical outcomes, necessitating a gold-standard diagnostic framework for precise phenotyping.

The nasal allergen provocation test (NAPT), internationally recognized as the diagnostic gold standard for AR and local allergic rhinitis, directly applies allergens to nasal mucosa to elicit or exacerbate symptoms. Endorsed by global guidelines (e.g., ARIA, EPOS), NAPT has demonstrated safety through over a decade of clinical refinement. Despite its advantages, current protocols involve multi-dose allergen challenges at varying concentrations, rendering the procedure time-prohibitive and limiting clinical adoption. Developing a simplified, standardized provocation method is an urgent unmet need to expedite practical application.

ELIGIBILITY:
Inclusion Criteria:

AR patients:

* Aged 18-75 years;
* patients who visited the Department of Otorhinolaryngology,the First Affiliated Hospital of Nanjing Medical Uncversity and were willing to undergo nasal provocation test; 3.Ptients who are willing to provide specimens for free to promote the study of the diagnostic efficacy of nasal provocation.

Healthy volunteers:

* Aged 18-75 years;
* Did not have any nasal symptoms and tested negative for allergens

Exclusion Criteria:

* Acute rhinosinusitis or acute exacerbation of chronic rhinosinusitis; active phase or symptom exacerbation of allergic diseases (e.g., allergic rhinitis, asthma).
* History of severe allergic reactions (e.g., anaphylaxis).
* Severe chronic obstructive pulmonary disease (COPD) or severe cardiopulmonary diseases contraindicating epinephrine use.
* Active phase of other severe systemic diseases (e.g., malignancies, autoimmune diseases).
* Within 1 week post-vaccination.
* Pregnancy, lactation, or preconception period.
* Inability to comply with study procedures (particularly children under 5 years old).
* Recent nasal surgery (within 2 months), nasal deformities (e.g., choanal atresia, severe nasal septum deviation/perforation), dry/atrophic rhinitis, severe nasal obstruction (e.g., hypertrophic rhinitis, rhinitis medicamentosa), or uncontrolled epistaxis.
* Current use of anti-allergy medications, including:Intranasal agents: corticosteroids, antihistamines, decongestants, anticholinergics, sodium cromoglicate;Systemic agents: oral antihistamines, oral/injectable corticosteroids.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1.Aged 18-75 years; 2. patients who visited the Department of Otorhinolaryngology,the First Affiliated Hospital of Nanjing Medical Uncversity and were willing to undergo nasal provocation test; 3.Ptients who are willing to provide specimens for free to promote the study of the diagnostic efficacy of nasal provocation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale for nasal symptoms | The questionnaire should be done within 15 minutes after the nasal provocation test.
  Patients are scored by questionnaire before and after treatment, and the change in score before and after treatment is the primary outcome measure ,the value of the total scores change from 0 point to 40, higher scores mean a comparatively more positive outcome, which means the patient has a more severe symptoms.
total nasal symptom scores | The questionnaire should be done within 15 minutes after the nasal provocation test.
  Patients are scored by questionnaire before and after treatment, and the change in score before and after treatment is the primary outcome measure ,the value of the total scores change from 0 point to 12, higher scores mean a comparatively more positive outcome, which means the patient has a more severe symptoms.
4-phase rhinomanometry (4PR) measurements of nasal resistance | The measurements should be done within 15 minutes after the nasal provocation test.
  To measure the nasal resistance changes at 150Pa before and after the nasal provocation tests.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Cheng, PhD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
All the individual participant data only available to reasearchers participated in this study